CLINICAL TRIAL: NCT02373995
Title: Investigation of Novel Biomarkers and Definition of the Role of the Microbiome In Graves' Orbitopathy
Brief Title: Role of the Microbiome in Graves' Orbitopathy
Acronym: Indigo
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Cultech Ltd, Port Talbot, UK (Unknown); Universität Duisburg-Essen (Other); School of Medicine and School of Biosciences, Cardiff University, Cardiff, UK (Unknown); IDRA Laboratory, Parco Tecnologico Padano s.r.l, Lodi, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Indigo
Record Dates: First submitted 2015-01-29; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Graves' Disease
Keywords: Graves; Orbithopaty; euthyroidism; microbiome
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAB4 (Active Comparator): In addition to conventional Anti Thyroid Drug (ATD), LAB4 probiotic preparation will be administered at the 2 cps x 2/die dosing with food for 6 months. It is key to properly store LAB4 at 8°C.
  Interventions: Biological: LAB4
- Placebo (Placebo Comparator): In addition to conventional Anti Thyroid Drug (ATD) a LAB4 placebo preparation will be administered at the 2 cps x 2/die dosing with food for 6 months. It is key to properly store placebo at 8°C.

INTERVENTIONS:
Biological: LAB4 — Additional treatment with the specific LAB4 probiotic preparation
  Arms: LAB4

SUMMARY:
Graves' orbitopathy (GO), also known as thyroid eye disease, affects approximately 3 million people in Europe with an estimated socioeconomic burden of 6.4 billion euros per annum. GO is a complication of Graves' disease which is an autoimmune disease and the commonest cause of an overactive thyroid gland. The treatment of GO remains unsatisfactory and the majority of patients report long-term impairment of quality of life. The effects of gut derived antigens, from micro-organisms and nutrients, on the autoimmune response will be tested in the animal model by probiotic and "contra-biotic" intervention. In the Indigo interventional trial the investigators will add to the standard anti-thyroid drug treatment (ATD) a specifically designed probiotics (LAB4, Cultech Ltd., West Glamorgan, UK) to assess whether it is possible to modify the microbiome in GD patients and improve their immunological status.

DETAILED DESCRIPTION:
Investigation of Novel biomakers and Definition of the role of the microbiome In Graves' Orbitopathy (GO) (INDIGO)

Background Graves' orbitopathy (GO), also known as thyroid eye disease, affects approximately 3 million people in Europe with an estimated socioeconomic burden of 6.4 billion euros per annum. GO is a complication of Graves' disease which is an autoimmune disease and the commonest cause of an overactive thyroid gland. The treatment of GO remains unsatisfactory and the majority of patients report long-term impairment of quality of life. To improve the outcomes of people with GO and thus reduce long-term illness and cost to society, research is needed to address the identification of risk factors, develop a better understanding of the pathophysiology of the disease, devise approaches for early diagnosis during the pre-clinical stage of the disease, and create novel and safe interventions. The effects of gut derived antigens, from micro-organisms and nutrients, on the autoimmune response will be tested in the animal model by probiotic and "contra-biotic" intervention. In the Indigo interventional trial the investigators will add to the standard anti-thyroid drug treatment (ATD) a specifically designed probiotics (LAB4, Cultech Ltd., West Glamorgan, UK) to assess whether it is possible to modify the microbiome in GD patients and improve their immunological status.

Primary objective:

To modify the microbiome in GD patients to reduce pathogenic species and enrich its commensal, symbiotic components.

Secondary objective:

To decrease the anti-TSHr antibody titer and the concentration of IgG and IgA in GD patients.

Experimental design The investigators are interested in inducing potential modifications of the gut microbioma and in obtaining a reduction of the anti-THSr antibody titer and of the total IgG and IgA concentrations, so as to prevent relapse and development or progression of eye disease. In particular, the expected, beneficial modification of the gut microbioma relates to a reduction at the end of treatment of at least 5% of the Firmicutes:Bacteroides ratio and 30% of the anti-TSHr antibody titer and of total IgG and IgA concentrations.

Patients with a diagnosis of Graves' disease with or without OB will be randomized to receive either ATD plus LAB4 or ATD plus placebo for 6 months. LAB4 consists of 4 strains:

Lactobacillus acidophilus CUL21 (NCIMB 30156) Lactobacillus acidophilus CUL60 (NCIMB 30157) Bifidobacterium bifidum CUL20 (NCIMB 30153) Bifidobacterium animalis subsp. lactis CUL34 (NCIMB 30172) and will be administered orally, twice a day during meals, for 6 months. Samples of blood (for serum and DNA)and, tears (Schirmer strips), nasal swabs and faeces will be collected at the first visit, before any treatment or within 4 weeks of anti-thyroid drug (ATD) therapy commenced by community physician. The same samples will be collected on the first occasion that euthyroidism has been restored on the usual block/replace or titration regimen used locally. The same samples will also be collected 6 months after cessation of treatment or at the point of relapse if that is sooner .

High through-put analysis of microRNA (miRNA) in serum and proteomic analyses of tears and serum will be used to search for biomarkers predictive of eye disease progression . In addition, antibody responses will be analyzed to identify if microbial or food derived antigens are involved in triggering disease or associated with GO progression . Moreover, 16S RNA gene sequencing will serve to characterize the patients microbiomes to assess whether this information can be used to develop diagnostics for individuals at risk of GD and then of developing GO .

ELIGIBILITY:
Inclusion Criteria:

* Group A: Untreated Graves' hyperthyroidism (or within 4 weeks of initiating ATD treatment)
* definition hyperthyroidism: TSH decreased, FT4 and /or FT3 increased
* definition Graves': diffusely enlarged thyroid gland either by palpation or echograpy, and/or homogeneous thyroid uptake at scintigraphy, or positive TSHRAb
* first episode or recurrence of Graves' hyperthyroidism
* minimal or no eye signs, defined as lid retraction / lid lag but no other signs.

Planned treatment with antithyroid drugs either titration regimen or block-and-replace regimen for 18 months.

Group B. Untreated Graves' hyperthyroidism (or within 4 weeks of initiating ATD treatment) with overt signs of GO as defined by EUGOGO1

1. Mild GO: patients whose features of GO have only a minor impact on daily life insufficient to justify immunosuppressive or surgical treatment. They usually have only one or more of the following: minor lid retraction (<2 mm), mild soft tissue involvement, exophthalmos <3 mm above normal for race and gender, transient or no diplopia, and corneal exposure responsive to lubricants)
2. Moderate-to-severe GO: Patients without sight-threatening GO whose eye disease has sufficient impact on daily life to justify the risks of immunosuppression (if active) or surgical intervention (if inactive). Patients with moderate-to-severe GO usually have any one or more of the following: lid retraction R2 mm, moderate or severe soft tissue involvement, exophthalmos >3 mm above normal for race and gender, inconstant, or constant diplopia.
3. Sight -threatening GO: Patients with dysthyroid optic neuropathy (DON) and/or corneal

Exclusion Criteria:

* Previous or planned treatment with 131I or thyroidectomy (A&B); sight threatening GO requiring decompression (B); drugs interfering with the natural course of GO (A&B): steroids, immunosuppressants, thiazolidinediones, antibiotics / antifungals / antivirals (both topical and systemic for at least 4 weeks prior to recruitment to the study); acute diarrhea illness (gastroenteritis for at least 4 weeks prior to recruitment to the study); Drugs interfering with thyroid function (A&B): amiodarone, lithium, iodine supplements; Drug or alcohol abuse (A&B); no informed consent (A&B); Age less than 18 (A&B); Pregnancy (A&B).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Microbiome modification (beneficial modification of the gut microbioma relates to a reduction at the end of treatment of at least 5% of the Firmicutes:Bacteroides ratio and 30% of the anti-TSHr antibody titer and of total IgG and IgA concentrations) | 6 months
  modification the microbiome in GD patients to reduce pathogenic species and enrich its commensal, symbiotic components. The proportion (%) of each species will be assessed and recorded.

SECONDARY OUTCOMES:
Improvement immunological status (antibody responses will be analyzed to identify if microbial or food derived antigens are involved in triggering disease or associated with GO progression) | 6 months
  To decrease the anti-TSHr antibody titer and the concentration of IgG and IgA in patients with Graves' disease. The concentration of each parameter will be assessed in mg/dl and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Salvi, MD, Principal Investigator — IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico Milano
Locations (1):
- Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Result] Bartalena L, Baldeschi L, Dickinson A, Eckstein A, Kendall-Taylor P, Marcocci C, Mourits M, Perros P, Boboridis K, Boschi A, Curro N, Daumerie C, Kahaly GJ, Krassas GE, Lane CM, Lazarus JH, Marino M, Nardi M, Neoh C, Orgiazzi J, Pearce S, Pinchera A, Pitz S, Salvi M, Sivelli P, Stahl M, von Arx G, Wiersinga WM; European Group on Graves' Orbitopathy (EUGOGO). Consensus statement of the European Group on Graves' orbitopathy (EUGOGO) on management of GO. Eur J Endocrinol. 2008 Mar;158(3):273-85. doi: 10.1530/EJE-07-0666. No abstract available. PMID 18299459